CLINICAL TRIAL: NCT03542721
Title: A Placebo-controlled, Randomized, Double-blind, Parallel, Multi-center Clinical Trial to Evaluate the Efficacy and Safety of DA-5515 (Circulan® Soft Cap.) in Patients With Chronic Fatigue Symptoms Due to Impaired Blood Circulation
Brief Title: Effect of DA-5515 (Circulan® Soft Cap.) in Patients With Chronic Fatigue Symptoms Due to Impaired Blood Circulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA-5515
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Fatigue Symptom
Keywords: chronic fatigue symptom; blood circulation
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo of DA-5515 Capsule (Placebo Comparator): Placebo of DA-5515 (three times a day)
  Interventions: Drug: Placebo of DA-5515
- DA-5515 Capsule (Experimental): Garlic oil, Gingko biloba ex.,Crataegus berry ex.,Melissa officinalis ex., (three times a day)
  Interventions: Drug: DA-5515

INTERVENTIONS:
Drug: DA-5515 — Crataegi ethanol extract, Garlic oil, Ginkgo leaf extract, Melissa folium extract (three times a day)
  Other Names: Circulan® Soft Capule
  Arms: DA-5515 Capsule
Drug: Placebo of DA-5515 — Placebo (three times a day)
  Other Names: Placebo capsule
  Arms: Placebo of DA-5515 Capsule

SUMMARY:
The aim of the present clinical study is to evaluate the efficacy and safety of the DA-5515 (Circulan Soft Cap.) in patients with chronic fatigue symptoms due to impaired blood circulation.

DETAILED DESCRIPTION:
This study is conducting to assess the efficacy and safety of the DA-5515 (Circulan Soft Cap.), which has been known to have a fatigue recovery effect due to impaired blood circulation.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford's category 0/0 or Ⅰ/1
* ABI <1.0
* CIS greater than 76
* HADS less than or equal to 10
* Subjects who have fatigue symptoms more than 1 month

Exclusion Criteria:

* Subjects who have diseases that can cause fatigue
* Subjects who are taking medication that can cause fatigue

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
CIS(Checklist Individual Strength) less than or equal to 76 | 8weeks
  Rate of subjects whose CIS score has improved less than or equal to 76 at 8weeks

CONTACTS AND LOCATIONS:
Overall Officials: WhanSeok Choi, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No